CLINICAL TRIAL: NCT05914025
Title: The Effect of a Brief Online Behavioral Activation Intervention by Activity Type
Brief Title: The Effect of a Brief Online Behavioral Activation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto University (Other)
Responsible Party: Principal Investigator, Parker Benson, Principal Investigator, Palo Alto University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-082
Record Dates: First submitted 2022-02-02; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Activation Intervention (Experimental): All individuals enrolled in the study will be assigned to this arm and will receive a brief behavioral activation psychoeducation module among other self-report assessments.
  Interventions: Behavioral: Behavioral Activation

INTERVENTIONS:
Behavioral: Behavioral Activation — Individuals will be provided with information about maladaptive patterns of behavior and how to correct these cycles with activity scheduling to elicit more positive emotional experiences. Participants will be provided with categories/lists of activities and a downloadable calendar after receiving the psychoeducation.

SUMMARY:
Depression is a worldwide phenomena that has a severe personal, social and societal impact. One such impact is an over $200 billion worldwide economic cost. While many treatments exist for depression, many individuals may not receive the support that they need for reasons such as stigma, financial restraints, or limited access to therapists. As such, it is important to assess the efficacy of brief online treatments as an alternative to full length, in-person treatments. A series of studies looking at a brief behavioral activation for depression treatment has shown that participants have reported temporarily improved mood, confidence, motivation and reduced depressive symptoms. It is important to test this treatment in multiple groups of people to acquire additional information regarding brief online interventions. This study seeks to collect participants from online social media sources and compare results to historical data that were collected from a prior research study which used Amazon Mechanical Turk as a recruitment source.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* United States Resident

Exclusion Criteria:

* Non-US resident
* Younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Depression level | 3 days
  Changes in depression score as measured by the PROMIS scale. The PROMIS is scored on a 5-point Likert scale with responses 1 to 5 corresponding to Never, Rarely, Sometimes, Often, and Always respectively.
Self-reported mood | 3 days
  Changes in mood as measured by a self-reported mood question. This measure is scored on a 9-point Likert scale (1 = Extremely Negative to 9 = Extremely Positive)
Daily Enjoyment | At time of original survey
  Changes in enjoyment as measured by a self-reported question around daily enjoyment. This measure is scored on a 5-point Likert scale (1 = Not at all to 9 = Extremely)

SECONDARY OUTCOMES:
Confidence, Motivation, and Usefulness | 3 days
  Changes in confidence, motivation, and usefulness are measured with single self-reported measures for confidence, motivation, and usefulness of the intervention. They are rated on a 9 point Likert scale (1 = Extremely Negative to 9 = Extremely Positive)

CONTACTS AND LOCATIONS:
Locations (1):
- Online Recruitment/Palo Alto University Campus, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No